CLINICAL TRIAL: NCT04908865
Title: A Multi-Center, Open-Label Study to Evaluate Safety, Efficacy and Pharmacokinetics of Belimumab Plus Standard Therapy in Chinese Paediatric Patients With Active Systemic Lupus Erythematosus (SLE)
Brief Title: Open-label Study of Belimumab Plus Standard Therapy in Chinese Pediatric Participants With Active Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213560
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Pediatric; Belimumab; Pharmacokinetics; Active Systemic Lupus Erythematosus; Safety; Efficacy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric participants receiving belimumab (Experimental)
  Interventions: Drug: Belimumab; Drug: Standard therapy

INTERVENTIONS:
Drug: Belimumab — Belimumab will be administered.
Drug: Standard therapy — Standard therapy will be continued.

SUMMARY:
This study will be conducted to evaluate the safety, efficacy and pharmacokinetics of belimumab administered in combination with background standard therapy in pediatric participants with active SLE.

ELIGIBILITY:
Inclusion criteria:

* Participants have or have had in series, 4 or more of the American College of Rheumatology (ACR) 11 criteria for the classification of SLE.
* Participant's age is 5 to 17 years at the time of informed consent.
* Have active SLE disease defined as a SELENA SLEDAI score >= 8 at screening (SELENA SLEDAI scoring).
* Have unequivocally positive autoantibody test results defined as an anti-nuclear antibody (ANA) titer >=1:80 and/or a positive anti-Double stranded deoxyribonucleic acid (dsDNA) serum antibody test.
* Are on a stable SLE therapy at Baseline. The stable treatment at Baseline consists of corticosteroids, anti-malarials, immunosuppressive/immunomodulatory agents and Non-steroidal anti-inflammatory drugs (NSAIDs), alone or in combination, at a fixed dose for a period of at least 30 days prior to Day 0.
* No gender restriction. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* The investigator, or a person designated by the investigator, will obtain written informed assent from each study participant or the participant's legally acceptable representative, parent(s), or legal guardian and the participant's assent, when applicable, before any study-specific activity is performed. The investigator will retain the original copy of each participant's signed assent document.

Exclusion Criteria:

* Have an estimated glomerular filtration rate (eGFR) as calculated by Schwartz Formula of less than 30 mL/minutes.
* Have acute severe nephritis defined as a significant worsening of renal disease (for example [e.g.], the presence of urinary sediments and other lab abnormalities) that, in the opinion of the study investigator, may lead to the participant requiring induction therapy with intravenous (IV) cyclophosphamide, Mycophenolate mofetil (MMF) or high dose corticosteroids during the first 6 months of the study.
* Have a history of a major organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Have clinical evidence of significant, unstable or uncontrolled, acute or chronic diseases not due to SLE (cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases) which, in the opinion of the investigator, could confound the results of the study or put the participant at undue risk.
* Have a planned surgical procedure or a history of any other medical disease (e.g., cardiopulmonary), laboratory abnormality, or condition (e.g., poor venous access) that, in the opinion of the investigator, makes the participant unsuitable for the study.
* Have a history of malignant neoplasm within the last 5 years.
* Have a history of a primary immunodeficiency.
* Have an Immunoglobulin A (IgA) deficiency (IgA level less than [<]10 mg/deciliters [milligrams/dL]).
* Have acute or chronic infections requiring management.
* Have recent infections that, in the opinions of the investigator, makes the participant unsuitable for the study or could put the participant at undue risk.
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 0.
* Have a Grade 3 or greater laboratory abnormality based on the protocol toxicity scale except for the following that are allowed:

  1. Stable Grade 3 prothrombin time (PT) secondary to warfarin treatment.
  2. Stable Grade 3 partial thromboplastin time (PTT) due to lupus anticoagulant and not related to liver disease or anti-coagulant therapy.
  3. Stable Grade 3 hypoalbuminemia due to lupus nephritis and not related to liver disease or malnutrition.
  4. Any grade proteinuria
  5. Stable Grade 3 gamma glutamyl transferase (GGT) elevation due to lupus hepatitis and not related to alcoholic liver disease, uncontrolled diabetes or viral hepatitis. If present, any abnormalities in the Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) must be Grade 2.
  6. Stable Grade 3 neutropenia; or stable Grade 3 lymphopenia; or stable Grade 3 leukopenia, due to SLE
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.
* Have evidence of serious suicide risk including any history of suicidal behavior in the last 6 months or who in the investigator's judgment, poses a significant suicide risk.
* Have received treatment with belimumab at any time.
* Have received any of the following within 364 days of Day 0:

  1. Treatment with any B-cell targeted
  2. Abatacept
  3. A biologic investigational agent
* Have required 3 or more courses of systemic corticosteroids for concomitant conditions (e.g., asthma, atopic dermatitis) within 90 days of Day 0.
* Have received any of the following within 90 days of Day 0:

  1. Anti-Tumour Necrosis Factor (TNF) or anti-interleukin (IL)-6 therapy (e.g., adalimumab, etanercept, infliximab, tocilizumab certolizumab, golimumab)
  2. Interleukin-1 receptor antagonist (anakinra)
  3. Intravenous immunoglobulin (IVIG)
  4. Plasmapheresis
* Have received any of the following within 30 days of Day 0:

  1. IV cyclophosphamide
  2. A non-biologic investigational agent (30 days window OR 5 half-lives, whichever is longer)
  3. Any new immunosuppressive/immunomodulatory agent, anti-malarial, NSAID
  4. High dose prednisone or equivalent (>1.5 mg/kilogram/day) or any intramuscular or intravenous steroid injection.
* Have received a live or live-attenuated vaccine within 30 days of Day 0.
* Have active central nervous system (CNS) lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident [CVA], cerebritis or CNS vasculitis) requiring therapeutic intervention within 60 days of Day 0.
* Have required renal replacement therapy (e.g., hemodialysis, peritoneal dialysis) within 90 days of Day 0 or be currently on renal replacement therapy.
* Participation in an interventional clinical study either concurrently or within 6 months of screening. Participation in an observational study may be permitted.
* Have a historically positive test or test positive at screening for Human immunodeficiency virus (HIV) antibody.
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest X-rays (posteroanterior) and a positive (not indeterminate) QuantiFERON-TB Gold Plus test.
* Hepatitis B: Serologic evidence of Hepatitis B (HB) infection defined as Hepatitis B surface antigen positive (HBsAg+) or Hepatitis B core antibody positive (HBcAb+).
* Hepatitis C: Positive test for Hepatitis C antibody at screening.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- China (9):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Suzhou
  - GSK Investigational Site, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Belimumab: Participants with active systemic lupus erythematosus (SLE) received belimumab at 10 milligrams per kilogram (mg/kg) body weight by intravenous (IV) infusion over a minimum of 1 hour on Days 0, 14, 28, and then every 28 days through Week 48 in combination with standard therapy.
Period: Overall Study
Arm/Group | Belimumab
Started | 67
Pharmacokinetic (PK) Population (PK population consisted of all the participants who received at least one dose of study treatment and for whom at least one post belimumab treatment PK sample was obtained and analyzed.) | 26
Completed | 59
Not Completed | 8
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 5
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Belimumab: Participants with active SLE received belimumab at 10 mg/kg body weight by IV infusion over a minimum of 1 hour on Days 0, 14, 28, and then every 28 days through Week 48 in combination with standard therapy.
Arm/Group | Belimumab
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 13.0 (2.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs) Through Week 52
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. AESIs included malignancies, post-infusion systemic or hypersensitivity reactions, infections (including serious infections of special interest), and depression, suicide, or self-injury. Infections of special interest included opportunistic infections (OI), herpes zoster (HZ), tuberculosis (TB), and sepsis. Number of participants with AESIs as identified by custom Medical Dictionary for Regulatory Activities (MedDRA) query has been reported.
Time Frame: Up to Week 52
Population: Intent-to-Treat (ITT) population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab
Number analyzed (Participants) | 67
Participants
  All malignancies | 0
  Post-infusion systemic reactions (PISR) | 0
  All infections of special interest (OI, HZ, TB, sepsis) | 2
  Depression (including mood disorders and anxiety)/suicide/self-injury | 0

2. Primary Outcome: Number of Participants With Greater Than Equal to (>=) 4 Points Reduction From Baseline to Week 52 in Safety of Estrogen in Lupus National Assessment - Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) Score
Description: The SELENA-SLEDAI score is a cumulative and weighted index for assessing SLE disease activity in participants with SLE. It consists of 24 disease descriptors related to signs and symptoms, laboratory tests, and physician's assessment across 9 organ systems. Each descriptor is assigned a weighted score (8 descriptors with a weight of 8 each, 6 descriptors with a weight of 4 each, 7 descriptors with a weight of 2 each, and 3 descriptors with a weight of 1 each) which is added up if the descriptor is observed during a visit or within the preceding 10 days. The total score ranges from 0 (no disease activity) to 105 (all 24 descriptors present simultaneously). A higher score indicates a more significant degree of disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Number of participants with a decrease of 4 points or more in the score at Week 52 compared to their Baseline score is presented.
Time Frame: Baseline (Day 0) and Week 52
Population: ITT population consisted of all participants who received at least one dose of study treatment. One participant with Baseline SELENA-SLEDAI score less than 4 was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab
Number analyzed (Participants) | 66
Participants | 44

3. Secondary Outcome: Number of Participants With AEs and Serious Adverse Events (SAEs) Through Week 52
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, is a birth defect or congenital anomaly, or other situations as per the medical or scientific judgment of the investigator. Number of participants with AEs and SAEs has been reported.
Time Frame: Up to Week 52
Population: ITT population consisted of all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Belimumab
Number analyzed (Participants) | 67
Participants
  AEs | 56
  SAEs | 19

4. Secondary Outcome: Percentage of Participants With >=4 Points Reduction From Baseline in SELENA-SLEDAI Score by Each Visit
Description: The SELENA-SLEDAI score is a cumulative and weighted index for assessing SLE disease activity in participants with SLE. It consists of 24 disease descriptors related to signs and symptoms, laboratory tests, and physician's assessment across 9 organ systems. Each descriptor is assigned a weighted score (8 descriptors with a weight of 8 each, 6 descriptors with a weight of 4 each, 7 descriptors with a weight of 2 each, and 3 descriptors with a weight of 1 each) which is added up if the descriptor is observed during a visit or within the preceding 10 days. The total score ranges from 0 (no disease activity) to 105 (all 24 descriptors present simultaneously). A higher score indicates a more significant degree of disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Percentage of participants with a decrease of 4 points or more in the score at each visit compared to their Baseline score is presented.
Time Frame: Baseline (Day 0) and Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: ITT population. 1 participant with Baseline SELENA-SLEDAI score below 4 was excluded. All 66 participants served as denominator to calculate percentages at each visit. For all visits except Week 52 (where percentage value was rounded off as no data was missing), missing data from missed visits were handled by multiple imputation. Estimates generated for every imputed dataset were combined by Rubin's rules to obtain percentages. So reported percentages may not yield whole number of participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Belimumab
Number analyzed (Participants) | 66
Percentage of Participants
  Week 4 | 39.8
  Week 8 | 51.8
  Week 12 | 68.9
  Week 16 | 69.0
  Week 20 | 65.4
  Week 24 | 68.1
  Week 28 | 65.7
  Week 32 | 67.7
  Week 36 | 69.1
  Week 40 | 75.1
  Week 44 | 74.2
  Week 48 | 71.3
  Week 52 | 66.7

5. Secondary Outcome: Change From Baseline to Week 52 in Physician Global Assessment (PGA)
Description: The PGA is used to assess the participant's current disease activity by investigator. It is collected on a 10 centimeter (cm) visual analogue scale. The score ranges from 0 (no activity) to 3 (severe activity). Lower score means no disease activity, higher score means severe disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 0) and Week 52
Population: ITT population consisted of all participants who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Belimumab
Number analyzed (Participants) | 67
Scores on scale | -0.931 (0.6046)

6. Secondary Outcome: Change From Baseline to Week 52 in Parent Global Assessment (ParentGA)
Description: The ParentGA is used to assess the participant's overall well-being at the moment rated on a 21-numbered circle visual analog scale by the parent. The score ranges from 0 (very well) to 10 (very poorly). Higher score indicates worse effect of the illness on the child. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 0) and Week 52
Population: ITT population consisted of all participants who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Belimumab
Number analyzed (Participants) | 67
Scores on scale | -2.71 (2.713)

7. Secondary Outcome: Change From Baseline in Average Daily Prednisone Equivalent Dose at Week 52
Description: The average daily prednisone equivalent dose accounted for all steroids taken IV, intramuscularly (IM), subcutaneously (SC), intradermally, and orally for both SLE and non-SLE reasons. All steroid dosages were converted to a prednisone equivalent in mg at each visit. The daily prednisone equivalent dose for a steroid was calculated as follows: collected dose of the steroid in mg multiplied by (*) conversion factor * frequency factor. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. At Baseline, the average daily prednisone equivalent dose was the sum of all prednisone doses over 7 consecutive days up to but not including Day 0, divided by 7. The average daily prednisone dose at Week 52 visit was the sum of all prednisone doses over 7 consecutive days up to and including the Week 52 visit, divided by 7. Average daily prednisone equivalent dose was expressed in milligrams per day.
Time Frame: Baseline (Day 0) and Week 52
Population: ITT population consisted of all participants who received at least one dose of study treatment. 'Overall Number of Participants Analyzed' included only those participants who were analyzed (i.e., contributed data reported in table).
Measure: Mean (Standard Deviation); unit: milligrams per day
Arm/Group | Belimumab
Number analyzed (Participants) | 59
milligrams per day | -6.020 (9.2970)

8. Secondary Outcome: Time to First Flare Over 52 Weeks
Description: The SLE flare index (SFI) is used to categorize SLE flares as mild/moderate or severe. A mild/moderate SFI flare involves: a SELENA-SLEDAI score increase of 3 to 12 points (higher score means greater disease activity); SLE symptom development; prednisone dose increase (but not above 0.5 milligrams per kilogram per day [mg/kg/day]); non-steroidal anti-inflammatory drugs (NSAIDs)/hydroxychloroquine addition; or PGA score increase by 1 or more, but not to more than 2.5 (higher score means greater disease activity). A severe SFI flare involves: SELENA-SLEDAI score increase over 12 points; onset or worsening of severe SLE symptoms; prednisone dose increase above 0.5 mg/kg/day; introduction of potent immunosuppressants; hospitalization; or PGA score reaching 2.5 or higher. Time to first SLE flare (mild/moderate or severe) was the number of days from treatment start date until the participant met an event. Time to first flare was defined as event date minus treatment start date plus 1.
Time Frame: Up to Week 52
Population: ITT population consisted of all participants who received at least one dose of study treatment. 'Overall number of participants analyzed' included those participants who experienced a post-baseline SFI flare over 52 weeks.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Belimumab
Number analyzed (Participants) | 50
days | 141.0 [58.0 to 333.0]

9. Secondary Outcome: Time to First Severe Flare Over 52 Weeks
Description: The SFI is used to categorize SLE flares as mild/moderate or severe. A severe SFI flare involves SELENA-SLEDAI score increase over 12 points (higher score means greater disease activity), onset or worsening of severe SLE symptoms, prednisone dose increase above 0.5 mg/kg/day, introduction of potent immunosuppressants, hospitalization, or PGA score reaching 2.5 or higher (higher score means higher disease activity). Time to first severe SLE flare was the number of days from treatment start date until the participant met an event. Time to first severe flare was defined as event date minus treatment start date plus 1.
Time Frame: Up to Week 52
Population: ITT population consisted of all participants who received at least one dose of study treatment. 'Overall number of participants analyzed' included those participants who experienced a post-baseline severe SFI flare over 52 weeks.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Belimumab
Number analyzed (Participants) | 18
days | NA [289.0 to NA] — 'NA' indicates that the median time and/or interquartile range could not be estimated due to low number of events in the participants.

10. Secondary Outcome: Median Belimumab Concentration Levels at Day 0, 7, and 14 Days Post First Dose, and Pre-infusion and Post-infusion at Day 84
Description: Blood samples were collected at indicated time points for measurement of plasma concentrations of belimumab.
Time Frame: Days 0, 7, and 14 days post first dose, and pre-infusion and post-infusion at Day 84
Population: Pharmacokinetic (PK) population consisted of all the participants who received at least one dose of study treatment and for whom at least one post belimumab treatment PK sample was obtained and analyzed. 'Overall number of participants analyzed' included only those participants who were analyzed (i.e., contributed data reported in table). 'Number analyzed' included participants evaluable for specified time points.
Measure: Median (Full Range); unit: Micrograms per milliliter
Arm/Group | Belimumab
Number analyzed (Participants) | 26
Micrograms per milliliter
  Day 0: number analyzed (Participants) | 24
  Day 0 | 197.1173 [141.9326 to 257.3748]
  Day 7 | 71.3616 [35.9532 to 100.5913]
  Day 14 | 37.8585 [14.5944 to 74.1679]
  Day 84, pre-infusion: number analyzed (Participants) | 25
  Day 84, pre-infusion | 28.2415 [2.3467 to 89.0718]
  Day 84, post-infusion: number analyzed (Participants) | 25
  Day 84, post-infusion | 238.5688 [139.1862 to 357.0316]

11. Secondary Outcome: Apparent Total Clearance of Belimumab
Time Frame: Days 0, 7, and 14 days post first dose, and pre-infusion and post-infusion at Day 84
Reporting Status: Not Posted, anticipated posting 2026-06

12. Secondary Outcome: Volume of Distribution of Belimumab
Time Frame: Days 0, 7, and 14 days post first dose, and pre-infusion and post-infusion at Day 84
Reporting Status: Not Posted, anticipated posting 2026-06

13. Secondary Outcome: Terminal Half-life (t1/2) of Belimumab
Time Frame: Days 0, 7, and 14 days post first dose, and pre-infusion and post-infusion at Day 84
Reporting Status: Not Posted, anticipated posting 2026-06

14. Secondary Outcome: Estimated Maximum Concentration (Cmax) of Belimumab at Steady State
Time Frame: Days 0, 7, and 14 days post first dose, and pre-infusion and post-infusion at Day 84
Reporting Status: Not Posted, anticipated posting 2026-06

15. Secondary Outcome: Estimated Minimum Concentration (Cmin) of Belimumab at Steady State
Time Frame: Days 0, 7, and 14 days post first dose, and pre-infusion and post-infusion at Day 84
Reporting Status: Not Posted, anticipated posting 2026-06

16. Secondary Outcome: Estimated Average Concentration (Cavg) of Belimumab at Steady State
Time Frame: Days 0, 7, and 14 days post first dose, and pre-infusion and post-infusion at Day 84
Reporting Status: Not Posted, anticipated posting 2026-06

17. Secondary Outcome: Area Under Plasma Concentration-time Curve (AUC) of Belimumab at Steady State
Time Frame: Days 0, 7, and 14 days post first dose, and pre-infusion and post-infusion at Day 84
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs, and non-serious adverse events (non-SAEs) were collected from the start of the study intervention (Day 0) up to the post-treatment follow-up visit at Week 64
Description: All-cause mortality, SAEs, and non-SAEs were reported for ITT population that comprised of all participants who received at least 1 dose of study treatment.
Arm/Group | Belimumab
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 20/67
Other Adverse Events (participants affected / at risk) | 57/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab (N=67)
Bronchitis (Infections and infestations) | 3 (3)
COVID-19 (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
H1N1 influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Myocarditis (Cardiac disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1)
Neuromyelitis optica spectrum disorder (Nervous system disorders) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belimumab (N=67)
Upper respiratory tract infection (Infections and infestations) | 31 (63)
COVID-19 (Infections and infestations) | 9 (9)
Coronavirus pneumonia (Infections and infestations) | 11 (11)
Bronchitis (Infections and infestations) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (13)
Hepatic function abnormal (Hepatobiliary disorders) | 9 (13)
Lymphocyte count decreased (Investigations) | 5 (9)
White blood cell count decreased (Investigations) | 4 (11)
Pyrexia (General disorders) | 7 (9)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Renal failure (Renal and urinary disorders) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Conjunctivitis (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Oral candidiasis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 2 (2)
Tinea versicolour (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Abscess soft tissue (Infections and infestations) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Herpangina (Infections and infestations) | 1 (1)
Mumps (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Face oedema (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 1 (1)
Intraocular pressure increased (Investigations) | 3 (3)
Neutrophil count increased (Investigations) | 2 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Blood immunoglobulin M decreased (Investigations) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1)
Bone density decreased (Investigations) | 1 (1)
CD19 lymphocytes decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Reticulocyte count increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1)
Xerophthalmia (Eye disorders) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Eyelid oedema (Eye disorders) | 1 (1)
Ocular hypertension (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Myocardial injury (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Endocrine hypertension (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Data has not been disclosed for PK parameters derived from population PK analysis, as this analysis, integrating data from Study 213560 and other studies, is still under discussion and review to fully understand the PK characteristics. The data for all pre-specified PK parameters will be disclosed by 30 June 2026.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT04908865/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT04908865/SAP_001.pdf